CLINICAL TRIAL: NCT01739660
Title: A Phase 1, Single Site, Open-Label Study to Assess the Pharmacokinetics (PK) and Pharmacodynamics (PD) of Pegloticase (KRYSTEXXA®) in Patients on Hemodialysis
Brief Title: Study to Assess Pegloticase (KRYSTEXXA®) in Patients on Hemodialysis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Savient Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: M0403; 10122 (Other: IND number)
Record Dates: First submitted 2012-11-29; First posted 2012-12-03 (Estimated); Last update posted 2013-10-25 (Estimated); Status verified 2013-10

CONDITIONS: Chronic Kidney Disease Stage 5
Keywords: Chronic Kidney Disease Stage 5; Hemodialysis; pegloticase
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Pegloticase

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Pegloticase (Experimental): Pegloticase 8 mg single intraveneous dose
  Interventions: Drug: Pegloticase

INTERVENTIONS:
Drug: Pegloticase — a single 8 mg iv (in the vein) dose before hemodialysis session
  Other Names: KRYSTEXXA

SUMMARY:
This is a Phase 1 single dose study conducted to evaluate the PK and PD of pegloticase administered to hemodialysis patients.

A single dose of pegloticase will be administered intravenously to male or female hemodialysis patients (N = 12) starting 3 hour prior to dialysis.

The study consists of a Screening Period, a Treatment Period, and Follow up Period.

DETAILED DESCRIPTION:
End stage renal disease (ESRD) patients that require hemodialysis typically undergo hemodialysis treatment 3 times per week. As such, medications can be dialyzed off, reducing their clinical effectiveness; this study is being conducted to understand how dialysis affects the pharmacokinetics (PK) and pharmacodynamics (PD) of pegloticase.

ELIGIBILITY:
Inclusion Criteria:

1. 18 and 75 years of age, inclusive
2. Agrees to employ best possible methods to abstain from becoming pregnant or impregnating another.
3. Stage V chronic kidney patients with minimal or no residual renal function receiving hemodialysis and stable on hemodialysis (3x week)
4. BMI = 18.5 kg/m2 to < 45 kg/m2

Exclusion Criteria:

1. Any surgical or medical condition that may interfere with drug absorption, distribution, metabolism, or excretion, or any other condition that may place the subject at risk

   1. Glucose-6-phosphate dehydrogenase (G6PD) deficiency
   2. Uncontrolled congestive heart failure
   3. Refractory chronic gout
2. History of drug and/or alcohol abuse within 6 months prior to screening
3. History of or current clinically significant mental disorder or an antagonistic personality that compromises the validity of the informed consent
4. Donation of blood or plasma within 30 days prior to dosing
5. History of or current hepatitis, or carriers of hepatitis B surface antigen (HbsAg) and/or hepatitis C antibodies (anti-HC).
6. Use of an investigational drug or product, within 30 days
7. History of clinically significant drug allergies or sensitivities
8. Females with a positive pregnancy test or who are breast feeding at Screening or plan to breast feed within 30 days of dosing
9. A baseline QTc interval ≥ 490 milliseconds for males and ≥ 510 milliseconds for females
10. Is unable to refrain from alcohol
11. Has taken any prescription or over the counter medication within 7 days prior to treatment day that, in the opinion of the Investigator, could be expected to confound the PK or metabolism of the study drug
12. Has taken the following herbal agents or nutraceuticals within 7 days prior to Screening: chapparal, comfrey, germander, gin bu huan, kava, pennyroyal, skullcap, St. John's Wort, or valerian
13. Has poorly controlled malignant hypertension (systolic blood pressure [SBP] > 200 mm Hg and/or diastolic blood pressure [DBP] > 120 mm Hg,
14. Concurrent use of urate-lowering drugs

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2012-12; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
• To evaluate the pharmacokinetics (PK) of pegloticase after a single-dose administration to hemodialysis patients when administered starting 3 hours before dialysis | 1 month

SECONDARY OUTCOMES:
• To evaluate the pharmacodynamics (PD) of pegloticase and SUA, before and after hemodialysis sessions | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Harry Alcorn, Pharm D, Principal Investigator — Davita Clinical Research
Locations (1):
- Davita Clinical Research, Minneapolis, Minnesota, United States